CLINICAL TRIAL: NCT04142606
Title: LUMIERE on the FETUS : A Study on the Added Value of Fetal MRI
Brief Title: LUMIERE on the FETUS
Acronym: FETUS
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: LUMIERE Fondation ( fondation-lumiere.org) under the aegis of Fondation de France (Unknown); University of Paris 5 - Rene Descartes (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190334
Record Dates: First submitted 2019-09-04; First posted 2019-10-29 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control Group (Group 1): Having prenatal ultrasound screening without detected abnormality
  Interventions: Other: fetal MRI
- Non Optimal Ultrasound Scan Group (Group 2): Having an ultrasound examination without abnormality detected but in whom ultrasound examination is not optimal (poor technical conditions, multiple pregnancies, obese patients)
  Interventions: Other: fetal MRI
- Malformation Group (Group 3): Standardized prenatal screening with ultrasound examination finding an isolated anomaly that does not currently constitute a commonly accepted indication of fetal MRI
  Interventions: Other: fetal MRI
- TOP Group (Group 4): A medical termination of pregnancy, (TOP), in addition to a fetopathological examination (virtopsy)
  Interventions: Other: fetal MRI

INTERVENTIONS:
Other: fetal MRI — The MRI examination added by this research, without injection or sedation, induces no risk for the mother as for the fetus (s)

SUMMARY:
Congenital anomalies are a major public health problem. They affect 2-3% of births, around 20,000 new cases per year in France, of which 15% are cared for in Ile de France. These congenital anomalies are a major cause of morbidity, infant mortality and disability. They are also a major cause of death during the infant period (22% of deaths during the first year of life: source CépiDC Inserm 2010). The detection, accurate diagnosis and accurate prognosis, particularly functional, of these congenital anomalies are still difficult in the current monitoring of pregnancy, which is based primarily on ultrasound. The use and development of modern imaging techniques is now essential to enable doctors to better see and better examine the fetus. Alongside ultrasound, Magnetic Resonance Imaging (MRI) is a technique that has undergone significant development in recent years. MRI must allow the effective anatomical and functional evaluation of the main fetal organs and could in particular be interesting in several situations in which it has not yet been sufficiently evaluated and is not yet performed in clinical routine.

DETAILED DESCRIPTION:
The inclusion will take place from 16WF to 36WG, within the framework of one of the 4 clinical subgroups of patients envisaged.

The standardized anatomic and functional MRI examination will in all cases last less than 45 minutes and will be based on sequences already used in clinical practice.

Clinical, biological, and ultrasound data will be collected prospectively and used for the usual management of the patient. For the purposes of the study, these data will be secondarily anonymized and analyzed in connection with the MRI data and the perinatal outcome to meet the specific objectives.

The lost-to-follow-up bias will be limited by the simplicity of the proposed perinatal surveillance, which does not differ from the surveillance usually recommended for these pregnancies

ELIGIBILITY:
Inclusion Criteria:

* patient ≥ 18 years
* Single or twin pregnancy
* gestational age≥ 16 WG and ≤ 36 WG based on cranio-caudal length (LCC) dating
* Collection of the patient's consent

Exclusion Criteria:

contraindication to MRI

* multiple pregnancies > 2
* subsequent follow-up impossible
* maternal condition contraindicates continuation of pregnancy
* patient having to have an MRI examination as part of the normal clinical follow-up of her pregnancy (identified or strongly suspected echocardiographic abnormality on ultrasound, diaphragmatic dome hernia, CMV fetal infection, antecedent brain abnormality in siblings, STT operated)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant patients followed in the Fetal Medicine Department of the Necker-Enfants Malades hospital belonging to one of the following 4 groups:
  * Having prenatal ultrasound screening without detected abnormality
  * Having an ultrasound examination without abnormality detected but in whom ultrasound examination is not optimal (poor technical conditions, multiple pregnancies, obese patients)
  * Standardized prenatal screening with ultrasound examination finding an isolated anomaly that does not currently constitute a commonly accepted indication of fetal MRI
  * A medical termination of pregnancy, in addition to a fetopathological examination (virtopsy)
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-12-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
feasibility of advanced MRI techniques | From inclusion to end of neonatal period (max 25 weeks)
  % of satisfactory sequences
feasibility of advanced MRI techniques | From inclusion to end of neonatal period (max 25 weeks)
  quality of standardized morphological fetal examination using recognizable criteria of normality
feasibility of advanced MRI techniques | From inclusion to end of neonatal period (max 25 weeks)
  quality of standardized functional fetal examination using recognizable criteria of normality

SECONDARY OUTCOMES:
concordance of information collected by MRI | From inclusion to end of neonatal period (max 25 weeks)
  Concordance of the diagnosis carried out on each standardized section in ultrasound, MRI and the final diagnosis: Standardized cuts with main anatomical landmarks seen and of usual appearance.
concordance of information collected by MRI | From inclusion to end of neonatal period (max 25 weeks)
  Concordance of the diagnosis carried out on each standardized section in ultrasound, MRI and the final diagnosis: Standardized cuts with main anatomical landmarks seen and unusual appearance.
Concordance of information collected by MRI | From inclusion to end of neonatal period (max 25 weeks)
  Concordance of the diagnosis carried out on each standardized section in ultrasound, MRI and the final diagnosis: Standardized cuts with main non-evaluable anatomical landmarks.
Acceptability of the examination for the patient: leackertLikert scale | Through MRI study completion an average of 6 months
  will be assessed by a Likert scale. which is a psychometric tool for measuring an attitude in individuals. It consists of one or more statements (statements or items) for which the respondent expresses her degree of agreement or disagreement (5 items from 1 to 5 points : from "very poor", "poor", "average", "good", "very good"). A scale of several items can be summarized by the average of the item scores.
Reproducibility of the examination analysis | After study completion, an average of one year
  will be assessed by means of Kappa coefficient
relevance of MRI | From inclusion to end of neonatal period (max 25 weeks)
  will be assessed by the % of added informations
Specific Absorption Rate for each type of sequence | After study completion, an average of one year
  SAR is an MRI machine parameter
feasibility of fusion imaging (echo / MRI) | After study completion, an average of one year
  will be assessed by the success rate of appropriate matching - % of successful echo-IRM fusion
norms of growth of main organs and placenta | After study completion, an average of one year
  Creating of normal curves by MRI measurements for length at various gestational ages
norms of growth of main organs and placenta | After study completion, an average of one year
  Creating of normal curves by MRI measurements: for width at various gestational ages
norms of growth of main organs and placenta | After study completion, an average of one year
  Creating of normal curves by MRI measurements for height at various gestational ages
norms of growth of main organs and placenta | After study completion, an average of one year
  Creating of normal curves by MRI measurements for volumes at various gestational ages
Establishment of an anatomical and functional database on a large group of healthy fetuses | After study completion, an average of one year
  Build up of normal atlas of MRI images in normal fetuses. We will stored anonymous images of fetal brain acquired thought gestation and anatomical and using functionnal sequences
Establishment of an anatomical and functional database on a large group of healthy fetuses | After study completion, an average of one year
  Build up of normal atlas of MRI images in normal fetuses. We will stored anonymous images of fetal thorax acquired thought gestation and anatomical and using functionnal sequences
Establishment of an anatomical and functional database on a large group of healthy fetuses | After study completion, an average of one year
  Build up of normal atlas of MRI images in normal fetuses. We will stored anonymous images of fetal heart acquired thought gestation and anatomical and using functionnal sequences
Establishment of an anatomical and functional database on a large group of healthy fetuses | After study completion, an average of one year
  Build up of normal atlas of MRI images in normal fetuses. We will stored anonymous images of fetal abdomen acquired thought gestation and anatomical and using functionnal sequences
Establishment of an anatomical and functional database on a large group of healthy fetuses | After study completion, an average of one year
  Build up of normal atlas of MRI images in normal fetuses. We will stored anonymous images of fetal limb acquired thought gestation and anatomical and using functionnal sequences
Establishment of an anatomical and functional database on a large group of healthy fetuses | After study completion, an average of one year
  Build up of normal atlas of MRI images in normal fetuses. We will stored anonymous images of placenta acquired thought gestation and anatomical and using functionnal sequences
Concordance of diagnosis | Termination of pregnancy (max 25 weeks)
  Concordance of diagnosis between virtual autopsy and foetopathology

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Salomon, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Necker - Enfants Malades Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bouachba A, Bartin R, De Jesus Neves J, Bussieres L, Grevent D, Virfollet J, Gauchard G, Bobet L, Roux N, Glemain B, Salomon LJ, Gorincour G. Normative range of MRI-based fetal body volume and association with ultrasonographically estimated fetal weight at 16-36 weeks: prospective study. Ultrasound Obstet Gynecol. 2025 Jul;66(1):81-88. doi: 10.1002/uog.29234. Epub 2025 May 26. PMID 40418192
- [Derived] Bartin R, Melbourne A, Bobet L, Gauchard G, Menneglier A, Grevent D, Bussieres L, Siauve N, Salomon LJ. Static and dynamic responses to hyperoxia of normal placenta across gestation with T2*-weighted MRI sequences. Ultrasound Obstet Gynecol. 2024 Aug;64(2):236-244. doi: 10.1002/uog.27609. PMID 38348601